CLINICAL TRIAL: NCT01332539
Title: An Observational Study to Assess the Burden of Drug-resistant Partial Epilepsy in Italy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114872
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-04

CONDITIONS: Epilepsy, Partial
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- drug-resistant partial epilepsy
  Interventions: Other: no intervention
- controlled partial epilepsy
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — non-interventional study
  Other Names: non-interventional study

SUMMARY:
observational, non-interventional study in 120 patients with drug-resistant partial epilepsy, comprising two phases: a 3-month retrospective and a 6-month prospective. As control group, 120 patients with controlled partial epilepsy will be enrolled. The objective of the study is to describe the burden of illness in this epileptic population both in terms of costs and of quality of life. Costs and quality of life will be also compared between the two populations.

DETAILED DESCRIPTION:
observational, non-interventional study in 120 patients with drug-resistant partial epilepsy, comprising two phases: a 3-month retrospective and a 6-month prospective.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Diagnosis of partial epilepsy, defined as active, drug-resistant in accordance to the 2010 ILAE (International League Against Epilepsy) definition and actually taking an add-on therapeutic regimen.
* Able and willing to give the written informed consent (to be obtained before any study assessment)

For each drug-resistant patient, will be enrolled a patient with the same diagnosis and actually taking an add-on therapy but with controlled epilepsy according to the 2010 ILAE definition.

Exclusion Criteria:

* Patient currently included in a clinical trial for an AED (Anti-Epileptic Drug)
* Hospital record data on epilepsy not available in the Investigator's files
* Patient unable to fill in self-questionnaires (quality of life instrument)
* Patient currently hospitalized
* Patient who, according to the Investigator's judgment, is not able to follow the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient with partial epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
total cost (direct and indirect) per patient per year of drug-resistant partial patients collected in the retrospective and in the prospective phase | 9 months: a 3-month retrospective and a 6-month prospective.

SECONDARY OUTCOMES:
The primary endpoint is the total cost (direct and indirect) per patient per year of controlled patients collected in the retrospective and in the prospective phase. | 9 months. a 3-month retrospective and a 6-month prospective.
the difference between the group of drug-resistant patients and the control group as regards each single resource consumptions and the direct and indirect costs (single and total) | 9 months: a 3-month retrospective and a 6-month prospective.
The comparison of the seven multi-item scores and the overall score of QOLIE-31 (Quality of life in Epilepsy -31 items) questionnaire between the two patients groups | questionnaire administerd at visit 1 only

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline